CLINICAL TRIAL: NCT05659875
Title: CompARing Long terM Outcomes in Chronic Stroke Survivors Across Investigational Assessments Following a Prescribed Upper Extremity Exercise Program (ARM-PROGRAM)
Brief Title: CompARing Long terM Outcomes in Chronic Stroke Survivors Across Investigational Assessments Following a Prescribed Upper Extremity Exercise Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Sean Savitz, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-22-0434
Record Dates: First submitted 2022-12-12; First posted 2022-12-21 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Chronic Stroke
Keywords: chronic stroke; stroke; arm impairment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARM-program (Experimental)
  Interventions: Other: Standard Occupational Therapy Arm Exercise Program

INTERVENTIONS:
Other: Standard Occupational Therapy Arm Exercise Program — Standard exercise program will be provided addressing shoulder, elbow, forearm, wrist, and hand with expectation that participant will complete 3 times a week. Exercise program will be updated at assessment timepoints as needed with change in arm function.
  Other Names: standard occupational therapy arm exercises

SUMMARY:
The purpose of the study is to compare assessments of arm function following a standard exercise program in chronic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Single qualifying stroke event as confirmed by CT or MRI
* At least 1 month post stroke
* Score of at least 2-/5 on Manual Muscle Test for wrist flexors or extensors, indicating adequate movement to complete robotic device use
* Able to follow written instructions

Exclusion Criteria:

* Prior arm injury impacting available passive or active range of motion or significant arm pain with movement
* Underlying brain pathologies such as metastatic or primary brain malignancies, comorbid multiple sclerosis, etc.
* Prior significant drug or alcohol abuse
* Diagnosed with dementia
* Pre-stroke baseline modified Rankin Scale (mRS) >3
* History of seizure/epilepsy
* History of clinically significant ischemic or hemorrhagic stroke prior to index stroke resulting in prior arm injury or weakness.
* Pregnancy
* Contraindication to MRI or Transcranial Magnetic Stimulation (TMS).
* Medical instability assessed by the treating stroke physician to participate to the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
change in arm impairment as assessed by Fugl Meyer - Upper Extremity assessment | Baseline, month 4, month 8, month 12, month 16, month 20, month 24
  This is a 33 item assessment and each is scored from 0 [unable to perform as instructed] - 2 [faultless performance] with a maximum score of 66. A higher number indicates better arm function.

SECONDARY OUTCOMES:
Change in integrity of corticospinal tract fibers as assessed by MRI with Diffusion Tensor Imaging (DTI). | Baseline, month 24
Change in motor evoked potential as assessed by Transcranial Magnetic Stimulation | Baseline, month 4, month 8, month 12, month 16, month 20, month 24

CONTACTS AND LOCATIONS:
Overall Officials: Sean Savitz, MD, Principal Investigator — UTHealth Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No